CLINICAL TRIAL: NCT07212335
Title: Single-Arm, Exploratory Clinical Study to Evaluate the Safety and Efficacy of Umbilical Cord Blood-Derived Mesenchymal Stem Cells in the Treatment of Long-Term Cytopenia After CAR-T Therapy
Brief Title: Safety and Efficacy of Umbilical Cord Blood-Derived Mesenchymal Stem Cells in the Treatment of Long-Term Cytopenia After CAR-T Therapy
Acronym: MSC-ICAHT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025028
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: Immune Effector Cell Associated Hematotoxicity
Keywords: ICAHT; hematotoxicity; CAR-T; cytopenia
MeSH Terms: conditions — Cytopenia

STUDY DESIGN:
Intervention Model Description: The study is divided into two phases: dose escalation phase and dose expansion phase.The dose escalation phase adopted a "3+3" design, with MTD (Maximum Tolerated Dose) determined by DLT (Dose-Limiting Toxicity) incidence. There are three groups: A, B, and C, with 3 subjects in each group. Group A: intravenous infusion of 2 × 10⁶ cells/kg body weight once; Group B: intravenous infusion of 2 × 10⁶ cells/kg body weight, once a week for 2 times; Group C: intravenous infusion of 2.0 × 10⁶ cells/kg body weight, once a week for 4 times. No DLT in three subjects means proceeding to the next higher dose group.One DLT in three subjects requires enrolling three more subjects.No DLT in these additions allows advancing to the higher dose group.The trial terminates when two or more DLTs occur in three or six subjects, with the current dose defined as MTD. In the dose expansion phase, investigators will select one specific dose test group (either A, B, or C) and expand the sample size by 6 subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC (Experimental): Mesenchymal stem cells: intravenous infusion, 2×10⁶ cells/kg body weight/week (once weekly), with 1 to 4 administrations based on different dosage groups.
  Interventions: Biological: Mesenchymal Stem Cell Infusion

INTERVENTIONS:
Biological: Mesenchymal Stem Cell Infusion — Mesenchymal stem cells: intravenous infusion, 2×10⁶ cells/kg body weight/week (once weekly), with 1 to 4 administrations based on different dosage groups.

SUMMARY:
This study is a single arm, open label, exploratory clinical study aimed at evaluating the efficacy, and safety of allogeneic umbilical cord blood-derived mesenchymal stem cells in the treatment of long-term cytopenia after CAR-T therapy.

DETAILED DESCRIPTION:
This is a single-center, open-label, dose-escalation exploratory trial, whose primary objective is to evaluate the safety and preliminary efficacy of human umbilical cord-derived mesenchymal stem cell injection in patients with acute lymphoblastic leukemia, lymphoma, and multiple myeloma who still suffer from severe cytopenia 3 weeks after CAR-T infusion, so as to provide dose evidence and efficacy reference for subsequent studies.

Targeting the severe cytopenia complication with a high incidence rate (27%-95%) after CAR-T therapy and limited efficacy of conventional treatments, this trial adopts a "3+3" dose-escalation design. All three groups use a unified single dose of 2×10⁶ cells/kg body weight, differing only in infusion frequency (Group A: once; Group B: twice; Group C: four times), with 3 patients initially enrolled in each group. The dose-limiting toxicity (DLT) observation period is 28 days; if 2 or more DLTs occur, dose escalation will be terminated. The total sample size ranges from 15 to 24 cases, with a 24-week follow-up (weekly for the first 8 weeks and monthly from week 9 to week 24).

Cell Preparation: Dispensed according to the actual body weight of each subject at a standard dose of 2×10⁶ cells/kg body weight, in compliance with GMP requirements. The cell viability is ≥85%, and the preparation can only be released after passing pathogenic microorganism, purity and tumorigenicity screenings.

Infusion Procedure: Administer 5mg dexamethasone 30 minutes before infusion to prevent allergies. Thaw and mix the preparation at room temperature before infusion, with an initial rate of 20 drops/min for the first 15 minutes; if no discomfort occurs, adjust the rate to 40-60 drops/min (completing the infusion within 30-60 minutes). Monitor vital signs every 15 minutes during infusion and keep the patient under observation for 2 hours after infusion.

Safety: Graded according to NCI CTCAE 5.0. Acute reactions are monitored for 24 hours, delayed reactions are specifically examined at weeks 4, 8, 12 and 24, and serious adverse events (SAEs) must be reported within 24 hours.

Efficacy: Complete response (CR) and partial response (PR) require "dual-test compliance + 7 days without blood product transfusion" (with an interval of ≥48 hours). The response rate and duration are calculated at weeks 4 and 8 as key time points.

Immunological Detection: Collect samples at baseline and at weeks 1, 4 and 8 after infusion to detect inflammatory markers, immune cells and cytokines.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all the following criteria to be enrolled in this study:

* 1.Voluntarily participate in the study and sign the informed consent form;
* 2.Aged ≥ 18 years, regardless of gender;
* 3.Patients with acute lymphoblastic leukemia (ALL), lymphoma, or myeloma who still have severe cytopenia (meeting any of the following conditions: absolute neutrophil count ≤ 1×10⁹/L; platelet count ≤ 30×10⁹/L; hemoglobin ≤ 70 g/dL) 3 weeks after CAR-T cell infusion;
* 4.ECOG performance status score ≤ 2;
* 5.Estimated survival time ≥ 6 months;
* 6.For female patients of childbearing potential, a negative pregnancy test result is required. Female patients of childbearing potential and male patients must use highly effective contraceptive measures during the study period and for 4 months/6 months after the discontinuation of treatment, respectively.

Exclusion Criteria

Patients with any of the following conditions are prohibited from enrolling in this study:

* 1.Having received other anti-tumor treatments (including but not limited to chemotherapy, radiotherapy, targeted therapy, immunotherapy, or hematopoietic stem cell transplantation) that may affect the hematopoietic system or blood cell count within 1 month before the screening period after CAR-T cell infusion;
* 2.Significant bone marrow infiltration by tumor cells during the screening period (for ALL: bone marrow morphological examination showing leukemia cell proportion > 5%; for multiple myeloma (MM) and lymphoma: bone marrow flow cytometry showing positive minimal residual disease (MRD), or bone marrow pathological immunohistochemistry showing lymphoma/clonal plasma cell infiltration);
* 3.Presence of any of the following conditions within 1 week before the first dose administration: infection with hemodynamic instability (requiring vasoactive drug support); deep fungal infection confirmed by imaging or microbiology (e.g., invasive aspergillosis, bloodstream infection, etc.); Pneumocystis jirovecii pneumonia, active tuberculosis, viremia (cytomegalovirus, parvovirus B19, etc.), and viral pneumonia (cytomegalovirus, COVID-19 virus, influenza virus, adenovirus, parainfluenza virus, etc.); as well as other severe infections that may affect hematopoiesis as judged by the investigator;
* 4.Serum creatinine or blood urea nitrogen ≥ 1.5 times the upper limit of normal (ULN);
* 5.Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 times ULN; total bilirubin ≥ 1.5 times ULN;
* 6.Other severe and/or uncontrolled diseases, or conditions that may affect study participation as judged by the investigator, including but not limited to: severe cardiac rhythm or conduction abnormalities (e.g., ventricular arrhythmias requiring clinical intervention, second-degree to third-degree atrioventricular block, etc.), corrected QT interval using Fridericia's formula (QTcF) > 480 ms on electrocardiogram; New York Heart Association (NYHA) heart function classification of Grade Ⅲ-Ⅳ; uncontrolled diabetes mellitus (glycated hemoglobin [HbA1c] > 9%); refractory hypertension; chronic obstructive pulmonary disease (forced expiratory volume in 1 second [FEV1] < 50% of predicted value), etc.;
* 7.History of arteriovenous thrombosis or atherosclerosis;
* 8.Positive for anti-human immunodeficiency virus (HIV) antibody or anti-Treponema pallidum specific antibody; positive for hepatitis B surface antigen (HBsAg); or positive for hepatitis B core antibody with hepatitis B virus deoxyribonucleic acid (HBV-DNA) > ULN; or hepatitis C virus ribonucleic acid (HCV-RNA) > ULN;
* 9.A history of or current malignant solid tumor (except cured non-invasive basal cell or squamous cell carcinoma of the skin and/or other cured carcinoma in situ; except other malignant tumors that have achieved clinical cure for > 5 years with no recurrence within 5 years);
* 10.Within 6 months after allogeneic hematopoietic stem cell transplantation, or donor cell chimerism rate ≤ 95%, or presence of active acute graft-versus-host disease (aGVHD) of Grade Ⅱ or higher, or moderate to severe chronic graft-versus-host disease (cGVHD);
* 11.Having received a live vaccine within 4 weeks before the first dose administration, or planning to receive any live vaccine during the study period;
* 12.Pregnant or lactating female patients;
* 13.Patients with mental disorders;
* 14.Participation in any other study drug trial (including vaccine trials) or exposure to other study drugs within 4 weeks or 5 half-lives (whichever is longer) before the first dose administration;
* 15.Patients who refuse to sign the informed consent form;
* 16.Other conditions deemed unsuitable for study inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From recruitment to 24 weeks after the last treatment.

SECONDARY OUTCOMES:
Complete Response (CR) rate | At Week 4 and Week 8 after the completion of MSC infusion
  Complete Response (CR) Criteria (no red blood cell/platelet transfusion for at least 7 days and meeting the standard in two consecutive tests):
  Hemoglobin (Hb) ≥ 100 g/L (for adults) or ≥ the lower limit of age-adjusted normal value; Absolute Neutrophil Count (ANC) ≥ 1.5×10⁹/L; Platelet Count (PLT) ≥ 100×10⁹/L.
Partial Response (PR) rate | At Week 4 and Week 8 after the completion of MSC infusion
  Partial Response (PR) Criteria: Meeting any of the following conditions (no red blood cell/platelet transfusion for at least 7 days and meeting the standard in two consecutive tests):
  Neutrophils: Absolute value increased by ≥ 0.5×10⁹/L compared with the baseline; Platelets: Absolute value increased by ≥ 10×10⁹/L compared with the baseline; Hemoglobin: Absolute value increased by ≥ 15 g/L compared with the baseline.
Overall Response (OR) rate | At Week 4 and Week 8 after the completion of MSC infusion
  OR=PR+CR
Response time | From the first MSC infusion to 8th week after the last MSC infusion
  The median time from the first MSC infusion to the first achievement of CR/PR for various blood cell types.
Duration of Relief（DOR） | from the date of achiving CR/PR to the earliest occurrence of hematopoietic indices falling below the CR/PR criteria or the end of the preset 24-week follow-up period after the first MSC infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences Hospital of Hematology (Chinese Academy of Medical Sciences Institute of Hematology), Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months to 36 months after study completion.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI